CLINICAL TRIAL: NCT02910570
Title: The Association Between Weight Loss With Subsequent Maintenance Using Liraglutide and Changes in Skin Autoflouresence in Overweight or Obese Patients With Knee Osteoarthritis - a Substudy to "Effect of Liraglutide on Body Weight and Pain in Overweight or Obese Patients With Knee Osteoarthritis: A Randomised, Double Blind, Placebo-controlled, Parallel Group, Single-centre Trial" (NCT02905864)
Brief Title: Changes in Skin Autoflouresence Following Weight Loss and Maintenance Using Liraglutide in Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Parker Research Institute (Other)
Responsible Party: Principal Investigator, Henrik Gudbergsen, MD, PhD, Parker Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 137.02
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide 3 mg (Experimental): Subjects will be up titrated to liraglutide 3 mg QD and stay on that dose for the remainder of the 52-week drug intervention period.
  Interventions: Drug: Liraglutide 3 mg (Saxenda)
- Liraglutide 3 mg placebo (Placebo Comparator): Subjects will be up titrated to liraglutide 3 mg placebo QD and stay on that dose for the remainder of the 52-week drug intervention period.
  Interventions: Drug: Liraglutide 3 mg placebo

INTERVENTIONS:
Drug: Liraglutide 3 mg (Saxenda) — Dose escalation scheme: Initial dosage of 0.6 mg per day, escalated bi-weekly by 0.6 mg to 3 mg per day over a total of 8 weeks
  Arms: Liraglutide 3 mg
Drug: Liraglutide 3 mg placebo — Dose escalation scheme: Initial dosage of a 0.6 mg drug equivalent volume per day, escalated bi-weekly by an 0.6 mg drug equivalent volume per day to a 3 mg drug equivalent volume per day over a total of 8 weeks.
  Arms: Liraglutide 3 mg placebo

SUMMARY:
This is sub-study to a randomised, double blind, placebo-controlled, parallel group, and single-centre trial investigating the effect of liraglutide on body weight and pain in overweight or obese patients with knee osteoarthritis (NCT02905864).

In the parent trial patients will be subjected to a run-in diet intervention phase (week -8 to 0) including a low-calorie diet and dietetic counselling. At week 0 patients will be randomised to receive either liraglutide 3 mg or liraglutide 3 mg placebo as an add-on to dietetic guidance on re-introducing regular foods and a focus on continued motivation to engage in a healthy lifestyle.

This sub-study of the parent trial only involves an additional assessment of skin auto fluorescence (AGE concentration) in the preallocation phase and in the main trial phase, i.e. from enrollment (defined as signature of informed consent) to treatment allocation (visits -Tx and T0 in the parent trial visit schedule) and from allocation to end of trial (visits T0 and T15 in the parent trial visit schedule).

ELIGIBILITY:
Same as parent trial (NCT02905864)

Inclusion Criteria:

* Informed consent obtained
* Clinical diagnosis of knee OA (American College of Rheumatology (ACR) criteria) confirmed by radiology but restricted to definite radiographic OA at early to moderate-stages (Kellgren-Lawrence grades 1, 2, or 3)
* Age ≥ 18 years and < 75 years
* Body mass index (BMI) ≥ 27 kg/m2
* Stable body weight during the previous 3 months (< 5 kg self-reported weight change)
* Motivated for weight loss

Exclusion Criteria:

* On-going participation, or participation within the last 3 months, in an organised weight loss programme (or within the last 3 months)
* Current or history of treatment with medications that may cause significant weight gain for at least 3 months before this trial
* Current use or use within three months before this trial of GLP-1 receptor agonist, pramlintide, sibutramine, orlistat, zonisamide, topiramate, or phentermine
* Type 1 diabetes
* Type 2 diabetes treated with glucose-lowering drugs other than metformin
* Alloplasty in target knee joint (see section 6.3)
* End stage disease in target knee joint (Kellgren-Lawrence grade 4)
* Immuno-inflammatory disease
* Chronic wide-spread pain
* Pregnancy or insufficient anti-conception therapy for female fertile patients
* Breast-feeding
* Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 x above upper normal range (UNR)
* Surgery scheduled for the trial duration period, except for minor surgical procedures
* Surgical procedures such as arthroscopy or injections into a knee within 3 months prior to enrolment
* Previous surgical treatment for obesity (excluding liposuction >1 year before trial entry)
* Thyroid stimulating hormone (TSH) outside of the range of 0.4-6.0 mIU/L
* Obesity secondary to endocrinologic or eating disorders or to treatment with medicinal products that may cause weight gain
* Family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2
* Inflammatory bowel disease
* Congestive heart failure, New York Heart Association (NYHA) class III-IV
* Diabetic gastroparesis
* History of or current diagnosis of pancreatitis (acute and/or chronic) or pancreatic cancer
* History of cancer with the exception of in-situ malignancies of the skin or cervix uteri
* History of major depressive disorder, a PHQ-9 (Patient Health Questionnaire-9) score of more than 15, or a history of other severe psychiatric disorders or diagnosis of an eating disorder
* Subjects with a lifetime history of a suicide attempt or history of any suicidal behaviour within the past month before entry into the trial
* Inability to speak Danish fluently
* A mental state impeding compliance with the program
* Use of opioids or similar strong analgesics
* Allergic reactions to the active ingredients of Saxenda, such as hypotension, palpitations, dyspnoea and oedema

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in advanced glycation end products in the skin | week 0 to 52
  advanced glycation end products levels will be measured on the skin of the volar side of the forearm using skin auto fluorescence

SECONDARY OUTCOMES:
Change in advanced glycation end products in the skin | week -8 to 0 (pre-randomisation weight loss intervention)
  advanced glycation end products levels will be measured on the skin of the volar side of the forearm using skin auto fluorescence.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik R Gudbergsen, MD, PhD, Principal Investigator — The Parker Institute
Locations (1):
- Department of Rheumatology, Frederiksberg, Capital Region, Denmark